CLINICAL TRIAL: NCT06900725
Title: Low-Dose Edoxaban Versus Very-Low-Dose Edoxaban in Elderly Patients With Atrial Fibrillation and a History of Stroke (LEAVE-Stroke): A Pragmatic Randomized Clinical Trial
Brief Title: Low Dose Edoxaban in Elderly Patients With AF and a History of Stroke
Acronym: LEAVE-Stroke
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University Hospital, Yun-Lin Branch (Other); National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202501081MINB
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Elderly; Atrial Fibrillation (AF); Ischemic Stroke
Keywords: very low-dose edoxaban; elderly; drug concentration; major bleeding; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke | interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LDER (Experimental): Patients will receive edoxaban 30 mg daily for stroke prevention.
  Interventions: Drug: Edoxaban 30 mg
- VLDER (Active Comparator): Patients will receive edoxaban 15 mg daily for stroke prevention.
  Interventions: Drug: edoxaban

INTERVENTIONS:
Drug: edoxaban — edoxaban 15 mg daily will be administered to the patients as secondary stroke prevention.
  Other Names: VLDER
  Arms: VLDER
Drug: Edoxaban 30 mg — edoxaban 30 mg daily will be administered to the patients as secondary stroke prevention.
  Other Names: LDER
  Arms: LDER

SUMMARY:
This prospectively enrolled, pragmatic randomized trial aims to investigate whether very low dose edoxaban regimen (15 mg daily) achieves similar edoxaban concentrations as low dose edoxaban regimen (30 mg daily), while maintaining a comparable risk of clinical outcomes and reducing major bleeding in elderly patients with atrial fibrillation and a history of ischemic stroke or transient ischemic attack.

DETAILED DESCRIPTION:
Edoxaban, a factor Xa inhibitor, is used to prevent stroke or systemic thromboembolism (SSE) in patients with atrial fibrillation (AF). In elderly patients, the post-hoc analysis of the Effective Anticoagulation with Factor Xa Next Generation in Atrial Fibrillation-Thrombolysis in Myocardial Infarction 48 (ENGAGE AF-TIMI 48) trial showed that a low-dose edoxaban regimen (LDER, 30 mg daily) reduced the risk of major bleeding compared to the standard-dose edoxaban regimen (SDER, 60 mg daily), without an offsetting increase in SSE risk. Furthermore, the Edoxaban Low-Dose for Elder Care Atrial Fibrillation Patients (ELDERCARE AF) trial demonstrated that a very-low-dose edoxaban regimen (VLDER, 15 mg daily) was more effective than placebo for elderly patients where standard anticoagulant intensity posed safety concerns. Although both LDER and VLDER appear suitable for the elderly population, data comparing these two regimens are lacking.

Specific purpose:

To investigate whether VLDER (15 mg daily) achieves similar edoxaban concentrations as LDER (30 mg daily), while maintaining a comparable risk of clinical outcomes and reducing major bleeding in elderly patients with AF and a history of ischemic stroke (IS) or transient ischemic attack (TIA) through a pragmatic randomized trial.

Study design:

The Very Low-Dose Edoxaban in Elderly Atrial Fibrillation Patients with a History of Stroke (LEAVE-Stroke) trial is a prospective, multicenter, randomized trial. Elderly patients aged ≥ 80 years with AF, a history of IS/TIA and concerns about the bleeding risk of standard anticoagulant intensity will be enrolled. Participants will be randomized to either the VLDER or LDER group.

Participant number: 120 patients (60 patients in each group). YEAR 1: Participant enrollment for the LEAVE-Stroke trial. YEAR 2: Continued participant enrollment, followed by a comparison of edoxaban concentration and clinical outcomes between two dose groups.

Study outcomes:

Primary outcome: The proportion of patients achieving edoxaban concentrations within the expected range from the ENGAGE-AF TIMI 48 trial (12-43 ng/mL at trough) at 1 month.

Secondary outcome: Major bleeding at 3 months, a composite of major bleeding, SSE or death at 3 months.

Significance: This pragmatic randomized trial will be the first to report real-world edoxaban concentrations in the VLDER group and to determine whether they are comparable to those in the LDER group. Furthermore, the study will provide insights into the short-term outcomes of VLDER in elderly patients with AF, a history of IS/TIA, and concerns about increased bleeding risk. These findings will not only inform edoxaban dosing strategies in clinical practice but also serve as a foundation for future large-scale, long-term studies to evaluate the feasibility and safety of using VLDER in this high-risk population.

Keywords: very low-dose edoxaban, elderly, drug concentration, major bleeding, atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Age>=80 years
* Has been diagnosed atrial fibrillation
* Has history of ischemic stroke or transient ischemic attack
* Has any of the bleeding risk lists below
* bodyweight < 60 kg
* creatinine clearance < 50 mL/min
* history of major bleeding or gastrointestinal bleeding
* concurrent use of antiplatelet agents (such as aspirin, clopidogrel, ticagrelor, prasugrel, cilostazol), non-steroidal anti-inflammatory drugs, amiodarone, tacrolimus, cyclosporine, dronedarone.

Exclusion Criteria:

* Has ever used anticoagulants, defined as:
* warfarin therapy within 1 month before study enrollment.
* using heparin, low molecular weight heparin or direct oral anticoagulants within 7 days before study enrollment.
* allergy to edoxaban
* under regular dialysis, includes hemodialysis or peritoneal dialysis
* refuse to provide informed consent.

Min Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving edoxaban concentrations within the expected range | 1 month
  The proportion of patients achieving edoxaban concentrations within the expected range from the ENGAGE-AF TIMI 48 trial (12-43 ng/mL at trough) at 1 month.

SECONDARY OUTCOMES:
Major bleeding | 3 months
  Major bleeding at 3 months
  Major bleeding is classified according to the Platelet Inhibition and Patient Outcomes (PLATO) criteria. Major life-threatening bleeding was defined as intracranial hemorrhage, intrapericardial bleeding, or overt bleeding leading to hemorrhagic shock, hypotension requiring inotropic agents or surgical intervention, or a hemoglobin reduction of more than 5 g/dL or necessitating a transfusion of ≥4 units of packed red blood cells. Other major bleeding events were classified as significant, disabling bleeding, or bleeding resulting in a hemoglobin decrease of 3-5 g/dL requiring a transfusion of 2-3 units of packed red blood cells.
Composite outcome | 3 months
  A composite of major bleeding, stroke or systemic thromboembolism or death.
  Stroke or systemic thromboembolism includes ischemic stroke (IS), transient ischemic attack (TIA), acute coronary syndrome, coronary artery disease, peripheral arterial occlusive disease, and venous thromboembolism.
  IS or TIA diagnoses were confirmed by brain computed tomography (CT) or magnetic resonance imaging (MRI). Brain CT angiography or perfusion was performed in patients with suspected large vessel occlusion. TIA was defined as a transient or reversible episode of neurological dysfunction lasting for < 24 h

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No